CLINICAL TRIAL: NCT03625648
Title: CSP #2008 - Pentoxifylline in Diabetic Kidney Disease
Brief Title: Pentoxifylline in Diabetic Kidney Disease
Acronym: PTXRx
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008
Record Dates: First submitted 2018-07-26; First posted 2018-08-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Kidney Disease
Keywords: Diabetic Kidney disease; pentoxifylline; PTX
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTX (Experimental): Active drug
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — The non-specific phosphodiesterase inhibitor pentoxifylline (PTX) was approved by the FDA in 1984 for the treatment of peripheral vascular disease.
  Arms: PTX
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Pentoxifylline (PTX) is a medication that has been on the market since 1984 for use in disease in the blood vessels of the legs. There is some preliminary information that it may protect the kidneys from damage due to diabetes and other diseases. "Pentoxifylline in Diabetic Kidney Disease" is a study to bee conducted in 40 VA hospitals across the nation to determine definitively whether or not PTX can prevent worsening of kidney disease and delay death in patients with diabetic kidney disease.

DETAILED DESCRIPTION:
Diabetic kidney disease (DKD) is the most frequent cause of chronic kidney disease (CKD) and end-stage renal disease (ESRD) in the U.S. and in U.S. Veterans. Control of blood pressure and reduction in proteinuria, for instance by blockade of the renin-angiotensin-aldosterone system (RAAS) with angiotensin-converting enzyme inhibitors (ACEIs) or angiotensin-receptors blockers (ARBs), have led to some improvement in outcomes in recent years. However, many patients continue to progress to ESRD, requiring costly dialysis or transplantation and resulting in high mortality. Patients with ESRD on maintenance dialysis also have markedly impaired quality of life. Thus, novel treatments are needed for this disease.

The non-specific phosphodiesterase inhibitor pentoxifylline (PTX) was approved by the FDA in 1984 for the treatment of peripheral vascular disease. Therefore, this drug has been in clinical use for over 3 decades and has been found to have an excellent safety profile. Recent experimental and clinical data suggest that PTX, when added to usual care in patients with DKD, leads to a reduction in albuminuria and reduced inflammation, as evidenced by lower levels of inflammatory cytokines, and may decrease progression of renal disease. The available evidence thus suggests the possibility of the use of PTX as a valuable repurposing of an old drug in the treatment of DKD. However, a large scale multicenter randomized clinical trial is needed to determine whether this agent can reduce hard endpoints such as ESRD and death in patients with DKD.

The objective of this study is to test the hypothesis that PTX, when added to usual care, leads to a reduction in the incidence of ESRD and mortality in type-2 diabetic patients with DKD when compared to usual care plus placebo.

The primary endpoint will be time to ESRD or death. ESRD will be defined as need for chronic dialysis or renal transplantation.

Secondary efficacy endpoints will be: (1) quality of life as measured by the Kidney Disease Quality of Life Short Form (KDQoL-SF), (2) time until doubling of serum creatinine, (3) hospitalization for congestive heart failure (CHF), (4) a three-point MACE (cardiovascular death, non-fatal myocardial infarction, non-fatal stroke), (5) peripheral vascular disease (PVD), (6) percentage of participants with 50% reduction in UACR from baseline, (7) Rate of change in eGFR per year during the study period. Safety (serious adverse events and adverse events possibly or probably related to study drug, discontinuation of study drug) will also be analyzed as a secondary safety outcome.

The design will be simple with only 2 face-to-face visits (randomization and end of trial visits). The remaining quarterly contacts can be conducted by telephone collecting minimal targeted information. Laboratory testing specifically for the study will be done only at randomization, at 6 months and the end of the study, if needed. However, coordinators will assure that a serum creatinine will have been measured every 6 months as part of routine clinical care or, in rare instances where one has not been done, obtain this measurement. Other than randomization to PTX or matched placebo, patient care will be handled by usual providers according to recommended standards of care.

There will be a one-year ramp-up phase which will include 6 VA hospitals. The purpose of the ramp-up phase will be to optimize procedures prior to widespread implementation, including assessing the recruitment rate to determine whether the expected rate can be achieved and assessing the efficacy of central distribution of study drug/placebo.

In addition, the investigators will refine methods of recruitment, demonstrate that the proposed follow-up methods are working as intended, and address unforeseen problems. This will be followed by the full study at 40 sites (which includes the 6 ramp-up sites) and will involve 3 years of recruitment and 5 years of follow-up.

Sample size calculation, assuming a 26.6% event rate in the control group and 21.6% event rate in PTX group (corresponding to a 19% relative reduction), two-sided alpha = 0.05, 85% power, a 3-year enrollment period, a minimum 5-year follow-up period, and one proposed interim analysis indicates that 2510 participants will need to be randomized.

If this study is successful and PTX is found to reduce the incidence of ESRD and/or death, this will reduce the personal and financial burden of renal replacement therapy (dialysis/transplantation) for Veterans with diabetic kidney disease

ELIGIBILITY:
Inclusion Criteria:

1. Type-2 diabetes.
2. Meet one of the following categories at a time that is greater than 90 days prior to randomization:

   * Group I: eGFR 15 to less than 30 mL/min/1.73 m2 regardless of the degree of albuminuria/proteinuria, or
   * Group II: eGFR 30 to less than 45 mL/min/1.73 m2 with UACR greater than or equal to (>) 30 mg/g or UPCR greater than or equal to (>) 150 mg/g, or
   * Group III: eGFR 45 to less than 60 mL/min/1.73 m2 with UACR greater than or equal to (>) 300 mg/g or UPCR greater than or equal to (>)500 mg/g
3. Participants need to be in one of the following categories at the time of randomization:

   * Group I: eGFR 15 to less than 30 mL/min/1.73 m2, or
   * Group II: eGFR 30 to less than 45 mL/min/1.73 m2 with UACR greater than or equal to (>) 30 mg/g, or
   * Group III: eGFR 45 to less than 60 mL/min/1.73 m2 with UACR greater than or equal to (>) 300 mg/g

Participants must be a United States Veteran, currently receiving care at a VA hospital with a local study team.

Exclusion Criteria:

1. Type 1 diabetes
2. History of non-diabetic kidney disease
3. Severe comorbid conditions expected to reduce life expectancy to less than 1 year, as determined by LSI
4. Active substance abuse, homelessness, or other condition that is likely to result in participant non,ompliance as determined by the LSI
5. Previous organ or bone marrow transplant
6. Pregnancy, breast feeding or female of child-bearing potential unwilling to use a reliable form of contraception
7. A recent (within 3 months) cerebral hemorrhage
8. Current use of oral pentoxifylline
9. Hypersensitivity to pentoxifylline or any of the components of the formulation
10. Current use of systemic ketorolac, oral or IV (contraindicated with pentoxifylline)
11. Current use of riociguat (contraindicated with pentoxifylline)
12. Current use of dialysis
13. Unable to provide informed consent
14. or any condition that in the opinion of the LSI would make the potential participant non-compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2376 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2028-01-03 (Estimated); Study Completion 2030-07-08 (Estimated)

PRIMARY OUTCOMES:
Time to ESRD or death | 5 to 9 years
  ESRD will be defined as need for chronic dialysis or renal transplantation.

SECONDARY OUTCOMES:
Quality of life (KDQoL-SF) | 5 to 9 years
  Quality of life as measured by the Kidney Disease Quality of Life Short Form (KDQoL-SF)
Time until doubling of serum creatinine | 5 to 9 years
  Time until doubling of serum creatinine
Incidence of congestive heart failure hospitalization (CHF) | 5 to 9 years
  The risk of a CHF hospitalization will be based on the participant-time data, specifically, the number of events per years.
Incidence of a three-point MACE | 5 to 9 years
  The risk of a MACE event will be based on participant-time data, specifically, the number of events per participant years.
Incidence of a peripheral vascular disease (PVD) | 5 to 9 years
  The risk of a PVD event will be based on participant-time data, specifically, the number of events per participant years.
Percentage of participants with 50% reduction in UACR from baseline | 5 to 9 years
  Percentage of participants with 50% reduction in UACR from baseline
Rate of change in eGFR per year during the study period | 5 to 9 years
  Rate of change in eGFR per year during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: David J Leehey, Study Chair — Edward Hines Jr. VA Hospital, Hines, IL
Locations (34):
- United States (34):
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, AR, Little Rock, Arkansas
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Harry S. Truman Memorial, Columbia, MO, Columbia, Missouri
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Leehey DJ, Carlson K, Reda DJ, Craig I, Clise C, Conner TA, Agarwal R, Kaufman JS, Anderson RJ, Lammie D, Huminik J, Polzin L, McBurney C, Huang GD, Emanuele NV. Pentoxifylline in diabetic kidney disease (VA PTXRx): protocol for a pragmatic randomised controlled trial. BMJ Open. 2021 Aug 16;11(8):e053019. doi: 10.1136/bmjopen-2021-053019. PMID 34400461